CLINICAL TRIAL: NCT02068898
Title: A Comparative, Proof of Concept Study, Comprising of a Pilot Phase Bioavailability Study Part and a Randomised, Cross-over Food-effect Study Part of "XS003" and Originator in Healthy Male Subjects
Brief Title: Pharmacokinetic Comparison of XS003 and Tasigna
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XSpray Microparticles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XS003_CT001
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- XS003 Dose-level 1 (Experimental): Capsule formulation
  Interventions: Drug: XS003
- XS003 Dose-level 2 (Experimental): Capsule formulation
  Interventions: Drug: XS003
- XS003 Dose-level 3 (Experimental): Capsule formulation
  Interventions: Drug: XS003
- Tasigna (Experimental): Marketed capsule
  Interventions: Drug: Tasigna

INTERVENTIONS:
Drug: XS003
  Other Names: RightSize Nilotinib
  Arms: XS003 Dose-level 1; XS003 Dose-level 2; XS003 Dose-level 3
Drug: Tasigna
  Other Names: Nilotinib
  Arms: Tasigna

SUMMARY:
The study will assess bioavailability of XS003 given as a single oral dose compared to Tasigna® given as a single oral dose in healthy male subjects.

DETAILED DESCRIPTION:
The study consists of two parts, the first part is composed as a pilot part and compares the bioavailability of single oral doses of XS003 compared to Tasigna® given as single oral dose in healthy male subjects. The second part is a food-effect part which assesses the food effect of a single oral dose of XS003 in healthy male subjects either fed or fasted. The study will also evaluate safety and tolerability of XS003 as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 18 to 55 years of age
* Body mass index (BMI) of 18.0 to 29.0 kg/m2
* Laboratory parameters in normal range

Exclusion Criteria:

* Females
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator.
* Subject has a QTcF>450 ms based on ECG at screening or a history of additional risk factors for Torsades de Pointe (e.g. hypokalaemia, hypomagnesemia, a family history of long QT syndrome)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Nilotinib | 3 days
  Pharmacokinetics measured by Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: XSpray Microparticles, Study Director — XSpray Microparticles
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom